CLINICAL TRIAL: NCT05131698
Title: Clinical Study of the Efficacy and Safety of Transhepatic Arterial Chemoembolization Combined With Tislelizumab and Lenvatinib in Patients With Advanced Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Zhi-ming Zhang, Chief Physician, Cancer Hospital of Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS2021（94）
Record Dates: First submitted 2021-11-04; First posted 2021-11-23 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Tislelizumab; Lenvatinib; TACE; Advanced Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — tislelizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with advanced unresectable liver cancer (Experimental)
  Interventions: Combination Product: Tislelizumab and Lenvatinib

INTERVENTIONS:
Combination Product: Tislelizumab and Lenvatinib — TACE therapy: For transarterial infusion chemotherapy before or after TACE embolization, each drug will generally be diluted with 0.9% sodium chloride solution or 5% dextrose solution 150-250 mL and injected slowly into the target artery for ≥20 min. Subsequent TACE therapy will be administered on an as-needed basis as assessed by the clinician, with each treatment interval exceeding 6 weeks and no more than 6 treatments in total.
  Lenvatinib: The starting dose of lenvatinib will depend on the patient's baseline weight: if baseline weight ≥ 60 kg, patients will receive 12 mg of lenvatinib administered once daily; if baseline weight < 60 kg, patients will receive 8 mg of lenvatinib once daily. TACE therapy will be given 3 days apart.
  Tirelizumab: Tirelizumab 200 mg , intravenous infusion on the same day as the first dose of lenvatinib, once every three weeks.
  Translated with www.DeepL.com/Translator (free version)
  Other Names: Clinical Study of the Efficacy and Safety of Transhepatic Arterial Chemoembolization Combined With Tislelizumab and Lenvatinib in Patients With Advanced Unresectable Hepatocellular Carcinoma

SUMMARY:
ICIs combined with AATDs have gradually become the mainstream treatment modality for advanced hepatocellular carcinoma, and more related clinical trials are underway. This is undoubtedly a breakthrough and the main direction for improving the overall 5-year survival rate of the liver cancer population in the next decade, and a touchstone for exploring the development and value of liver surgery in the era of comprehensive treatment for advanced hepatocellular carcinoma.

Overall, there are relatively few reports on various types of translational therapy for advanced HCC, probably for the following two reasons: (1) advanced hepatocellular carcinoma is complex, rapidly progressing, difficult to treat, and has low translational efficiency; (2) the existing translational therapy strategies are highly selective in terms of applicable population, complex treatment process, and institutional dependence, and cannot achieve efficient and successful translation.

At present, there are few studies reported on the application of TACE+ICIs+AATDs to carry out translational therapy. In the absence of relevant guidelines for reference, advanced hepatocellular carcinoma may be the best entrance to carry out translational therapy with ICIs combined with AATDs, and after satisfactory results are achieved in the treatment of this group of patients, a point-to-point effect can be generated, facilitating the transformation of TACE+ICIs+AATDs The target population of TACE+ICIs+AATDs translational therapy can be further expanded. To promote the development of hepatocellular carcinoma treatment and improve the long-term survival rate of the overall hepatocellular carcinoma population. In this study, we enrolled patients with advanced HCC and used TACE+ICIs+AATDs for conversion therapy to improve the conversion rate, so that unresectable HCC patients could be converted to a chronic disease state and achieve long-term survival on the one hand, and provide potential for sequential surgical treatment on the other. The drug of choice is lenvatinib. This study provides a basis for the clinical application of translational therapy for advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced Unresectable Hepatocellular Carcinoma
2. Histological examination or clinical diagnosis of HCC
3. BCLC C Stage
4. Child-Pugh A
5. ECOG 0-1
6. Age ≥ 18 years old and ≤ 70 years old
7. No serious concomitant diseases
8. No Portal vein tumor thrombus or Inferior vena cava tumor thrombus
9. No extrahepatic metastases
10. Not receiving any systematic treatment
11. life expectancy > 3 months.
12. The patient must be able to understand and be willing to sign a written informed consent form.

Exclusion Criteria:

1. previous (within 5 years) or concurrent other malignancies
2. participated in a clinical trial of another drug within four weeks
3. the presence of a contraindication to TACE
4. There is a history of bleeding, and any bleeding event with a severe grade of 3 or above in CTCAE v5.0 occurred within 4 weeks before screening
5. Patients with known CNS metastases or a history of CNS metastases prior to screening. For patients with clinically suspected CNS metastases, CT or MRI must be performed within 28 days prior to enrolment to exclude CNS metastases.
6. patients with a history of unstable angina pectoris; those with newly diagnosed angina pectoris within 3 months prior to screening or a myocardial infarction event within 6 months prior to screening; arrhythmias (including QTcF: ≥ 450 ms in men and ≥ 470 ms in women) requiring long-term antiarrhythmic medication and New York Heart Association classification ≥ Class II cardiac insufficiency.
7. Have a history of immunodeficiency, or suffer from other acquired and congenital immunodeficiency diseases, or have received allogeneic stem cell transplantation or organ transplantation in the past.
8. patients with infectious pneumonia, non-infectious pneumonia, interstitial pneumonia and other conditions requiring the use of corticosteroids.
9. Have a serious history of chronic autoimmune diseases, such as systemic lupus erythematosus. Well-controlled immune-related diseases, such as dermatitis, psoriasis and rheumatoid arthritis, can be included in the group after being evaluated by researchers.
10. There is a history of inflammatory bowel diseases such as ulcerative enteritis and Crohn's disease, and a history of inflammatory chronic diarrhea diseases such as irritable bowel syndrome.
11. Have a history of sarcoidosis or tuberculosis.
12. Known history of human immunodeficiency virus (HIV) infection.
13. patients with hypersensitivity to human or murine monoclonal antibodies.
14. persons with a history of psychotropic substance abuse who are unable to abstain or who have a psychiatric disorder.
15. patients with clinical signs of pleural effusion or peritoneal effusion requiring clinical intervention.
16. patients with concomitant illnesses that, in the judgment of the investigator, seriously jeopardize patient safety or interfere with patient completion of the study.
17. pregnant and lactating females.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-07-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 year
  Refers to cases in which the objective tumor outcome, including CR and PR, was assessed using the mRECIST version of the criteria

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi, China

REFERENCES:
- [Derived] Nong X, Yao Y, Xie J, Liang J, Zhang Y, Zhang Z. Preliminary experience of lenvatinib, tislelizumab and transcatheter arterial chemoembolization for BCLC stage C hepatocellular carcinoma: a phase II study. BMC Cancer. 2025 Oct 22;25(1):1631. doi: 10.1186/s12885-025-15016-9. PMID 41126100